CLINICAL TRIAL: NCT06039020
Title: ATGAM INTRAVENOUS INFUSION 250mg GENERAL INVESTIGATION
Brief Title: ATGAM General Investigation
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B5411004
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Aplastic Anemia
Keywords: ATGAM;; Anti-human thymocyte immunoglobulin, equine;; Aplastic anemia;
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anti-human thymocyte immunoglobulin, equine: Patients with moderate to severe aplastic anemia who receive ATGAM (Anti-human thymocyte immunoglobulin, equine)
  Interventions: Drug: Anti-human thymocyte immunoglobulin, equine

INTERVENTIONS:
Drug: Anti-human thymocyte immunoglobulin, equine — Usually, 40 mg of anti-human thymocyte immunoglobulin, equine per kilogram of body weight should be slowly administered by intravenous drip infusion once daily. The duration of treatment should be 4 days.

SUMMARY:
The objective of this study is to confirm the safety of ATGAM in patients with moderate to severe aplastic anemia under the actual use in Japan.

The registration criteria is patients with moderate to severe aplastic anemia who receive ATGAM.

The observation period is 24 weeks (6 months) from the start of administration (Day 1). However, in cases where treatment has been completed or discontinued less than 24 weeks after the start of administration, observation is continued until completion (discontinuation) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe aplastic anemia who receive ATGAM

Exclusion Criteria:

* No exclusion criteria is set out in this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe aplastic anemia who receive ATGAM
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse drug reactions (ADRs) | 24 weeks (6 months) from the start of administration (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5411004